CLINICAL TRIAL: NCT03933475
Title: A Feasibility Study of Telerehabilitation in East Riding for Patients With Cognitive Impairment Following Acquired Brain Injury
Brief Title: Telerehabilitation for Cognitive Impairment Following Acquired Brain Injury
Acronym: TRIER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hull University Teaching Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R2078
Record Dates: First submitted 2019-04-17; First posted 2019-05-01 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Cognitive Dysfunction; Brain Injuries
MeSH Terms: conditions — Cognitive Dysfunction; Brain Injuries

STUDY DESIGN:
Intervention Model Description: Pre and post intervention study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intendu Active Brain Trainer Telerehabilitation Games (Experimental): Use of telerehabilitation Games within the home environment
  Interventions: Device: Virtual reality game

INTERVENTIONS:
Device: Virtual reality game — Use of virtual reality games on television screens

SUMMARY:
Cognitive function is the mental action or process of acquiring knowledge and understanding through thought, experience, and the senses. Cognitive impairment describes a noticeable decline in cognitive function which can be temporary or permanent. This decline is measurable and ranges from mild to severe depending on the degree of decline in function. Cognitive impairment can be caused by a variety of diseases or conditions, and it is not limited to a specific age group. It can occur in patients following acquired brain injury such as traumatic brain injury and stroke. Some causes of cognitive impairment are related to health issues that may be treatable, such as medication side effects, vitamin B12 deficiency, and depression. Cognitive impairment has a significant impact on rehabilitation outcome and quality of life. It has significant health and economic impact. People with cognitive impairment report three times longer stay in hospital compared to people hospitalised for other conditions.

Cognitive rehabilitation is the process by which cognitive function can be improved and reduces the impact of cognitive impairment. Cognitive rehabilitation helps to improve functional outcomes and quality of life of patients with cognitive impairment. Current cognitive rehabilitation protocols use face to face interaction which cannot optimise the intensity of therapy due a lack of resources. Many areas of UK do not have dedicated cognitive rehabilitation service, programme or personnel and where it exists, the service is restricted largely to the urban centres. These services have high patient to staff ratio with prolonged waiting times often extending over 12 months to access input. Innovative technologies with telemedicine may well bridge the gap in service provision, improve engagement and offer opportunities in resource management.

Gamification refers to the application of typical elements of game playing (e.g. point scoring, competition with others, rules of play) to other areas of activity (such as healthcare) to encourage engagement and motivation. It is increasingly being used in rehabilitation and provides a means of developing more effective treatments and interventions. Practice and repetition are key rehabilitation processes that can be enhanced through the use of gamified innovative technology.

This protocol describes a trial of an innovative rehabilitation tool for community dwelling adults with cognitive impairment following acquired brain injury. The intervention is a novel interactive system connected to a television set using 3D cameras and tailored software to deliver therapeutic activities to patients within their homes. Each participant will be required to have 2 sessions per week using the device. Each session will last about 20 minutes with 4 different activities of 5 minutes duration each, targeting different domains of cognitive function. Follow up assessments will be carried out after 12 weeks of using the equipment.

The primary outcome measure will be the change in the assessment scores on the cognitive tests administered before and after undergoing the rehabilitation programme. Secondary outcomes on quality of life, participation in leisure time activities and satisfaction with the use of the equipment will also be obtained. Safety while using the device will be monitored and any side effects from engaging in the activities will also be monitored.

DETAILED DESCRIPTION:
The aim of the project is to explore the feasibility and effectiveness of using a telerehabilitation system to improve cognitive function in recruited study participants of community dwelling adult patients (over 18 years) with cognitive impairment secondary to acquired brain injury.

The study objectives are:

1. To investigate the feasibility through a pilot programme of utilising a telerehabilitation system to deliver cognitive rehabilitation to a cohort of East Yorkshire community dwelling patients within their home environment.
2. To investigate the feasibility that a cohort of community dwelling patients with post acquired brain injury cognitive impairment can participate in a 12-week duration therapy programme using a telerehabilitation system designed to improve domains of cognitive function (attention, reaction times, memory and executive function).
3. To investigate whether health related quality of life (HRQOL) is improved in study participants taking part in a 12-week programme of using a cognitive telerehabilitation system.
4. To investigate whether leisure time physical activity in increased in the study participants.

These study objectives will be achieved through measurement of the following outcome parameters:

1. Administering the Godin leisure time exercise questionnaire (Godin LTQ). This is a self-report paper-based questionnaire that will be administered pre and post intervention.
2. The HRQOL of patients with cognitive impairment following acquired brain injury as measured by the following self-report paper-based questionnaires: European quality of life -5 dimension (EQ-5D), fatigue severity scale (FSS) and the Short form 12 (SF-12). Mood will be assessed with the hospital anxiety and depression scale (HADS). These questionnaires will be administered pre and post intervention.
3. A user satisfaction questionnaire will be administered following the intervention as a measure of acceptance and satisfaction with engaging in guided self-rehabilitation through the use of telerehabilitation technology. This will be administered in the post intervention assessment only.
4. Baseline cognitive screening using the Montreal Cognitive Assessment (MoCA) test to determine suitability for the intervention.
5. Assessment of cognitive function of patients before and after the telerehabilitation intervention by administering the following questionnaires:

   1. Trail making and colour word interference subtests of the Delis-Kaplan Executive Function Systems (D-KEFS).
   2. Walking While Talking (WWT) - Executive Function test.
   3. The Repeatable Battery of the Assessment of Neuropsychological Status (RBANS). This is a screening measure that assesses: Immediate and delayed memory, Attention, Language and Visuospatial/Constructional skills.
   4. The Speed of Information Processing Subtests from the BIRT Memory and Information Processing Battery (BMIPB). This measures an individual's capacity for information processing, as well as their motor speed.

Study design The study design is a prospective pre-post intervention study aimed at evaluating cognitive rehabilitation in a sample of patients with cognitive impairment following acquired brain injury. The study primarily seeks to validate the feasibility of using purposefully designed videogames-based virtual reality technology to improve cognitive function in patients with cognitive dysfunction following acquired brain injury.

Recruited participants will undergo baseline assessments of cognitive function, leisure time activity, health related quality of life before engaging in a 12-week telerehabilitation programme using the Intendu functional brain trainer. Post intervention assessment using the same outcome measures administered in the baseline assessment will be performed 1 week after completion of the therapy programme.

The total duration of involvement for each participant is anticipated to be 14 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adults (>18 years)
* Clinical diagnosis of non-progressive Acquired brain injury cognitive Impairment.
* Must be able to stand independently for 20 minutes.
* Must be living in their own accommodation.
* Not involved in any ongoing clinical research.
* Must be able to communicate in English

Exclusion Criteria:

* Clinical diagnosis of photosensitive seizure disorders.
* Clinical diagnosis of Dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-10-31 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Cognitive Function: Memory, Attention, Language and Visuospatial skills | 6 months
  RBANS: The Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) provides a brief individually administered battery of tests to assess neuropsychological status and ideal for measuring change over time. It can be used to track recovery during rehabilitation. It is a 30-minute screening test comprising 12 subtests that assesses 5 domains: immediate and delayed memory, attention, language and visuospatial/constructional skills. Subtest raw scores are converted to age-based index scores. In addition, a total scale can be calculated. Reliability coefficients for assessment of change as well as test-retest reliability are high for the total scale.
Cognitive Function: Executive Function | 6 months
  DKEFS: The Delis-Kaplan Executive Function System (D-KEFS) measures verbal and non-verbal executive function in children and adults (ages 8-89 years). It comprises 9 tests each of which was designed as a standalone test. This study proposes to use some of the subtests namely; The Trail Making Test which measures flexibility of thinking on a visual-motor sequencing task and The Colour-Word Interference Test which measures ability to inhibit a dominant and automatic verbal response. The complexity of the tasks involved in administering the tests make them sensitive to the detection of even mild brain damage.
Cognitive Function: Divided Attention | 6 months
  WWT: The Walking While Talking test is a dual-task measure of divided attention to examine cognitive motor interactions. Variations of the WWT test exists and for this study, the test will be administered as follows:
  1. Walking - measure how many meters the participant walks, in 1 min (walk back and forth on a 10-meter section; instruct to turn around)
  2. Verbal fluency - while sitting down, count the number of words (excluding names and proper nouns), the participant says, beginning with a specific letter.
  3. Dual tasking - combine the two tasks. Measure how many words the participant says during 1 min, while walking. Note: use a different letter. Note: measure also the distance walked.
  The dual task motor cost (EF cost) is the difference in number of words generated between tests 2 and 3.
Cognitive Function: Information processing speed | 6 months
  Brain injury rehabilitation trust Memory and Information Processing Battery (BMIPB) is a group of tests used in assessing the effects of the damage to the brain on memory and speed of information processing (SoIP). It can assist in planning individual rehabilitation programmes and also in evaluating recovery. The SoIP test will be used from the BMIPB battery. On this test, the individual has to work through rows of five 2-digit numbers, cancelling the second highest number in each row. The task lasts 4 minutes. The individual then undertakes a 25 second motor speed cancellation task. Scores are expressed as percentiles. The difference between the scores obtained at initial testing and that obtained at retest are standardised and expressed as T scores. The test has high test- retest and interrater reliability. There is no significant floor or ceiling effects and practice effects are substantially eliminated through the use of different versions for test-retest.

SECONDARY OUTCOMES:
Health related quality of life (HRQOL) | 6 months
  EQ-5D-5L: The European Quality of Life Measure 5 Dimensions-5 Levels (EQ-5D-5L) is a standardised measure of health-related quality of life that can be used in a wide range of health conditions and treatments. It consists of a descriptive system and a visual analogue scale (EQ VAS). The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The scores on these five dimensions can be presented as a health profile or can be converted to a single summary index number. The EQ VAS records the patient's self-rated health on a vertical visual analogue scale. This can be used as a quantitative measure of health outcome that reflects the patient's own judgement.
Health related quality of life (HRQOL): Fatigue | 6 months
  FSS: The fatigue severity scale(FSS) is a 9-item tool that measures the severity of fatigue in a variety of conditions and its effects on an individual's activities and lifestyles. The FSS questionnaire comprises nine statements inquiring about the patient's usual way of life over the preceding week. Ratings are on a 7-point Likert scale, where higher scores indicate how strongly the patient agrees with the nine statements. A score of 36 and above (out of a maximum of 63) indicates the presence of significant fatigue. The FSS has been accepted as a simple and reliable measure of fatigue. This tool also incorporates the VAFS (visual analogue fatigue scale) on a horizontal visual analogue scale.
Health related quality of life (HRQOL): General health measure | 6 months
  SF-12: The SF-12 is a multipurpose short form (SF) generic measure of health status. 12-Item Short Form Health Survey (SF-12) was designed to reduce respondent burden while achieving minimum standards of precision for purposes of group comparisons involving multiple health dimensions. Two summary scores of health status, namely the physical component summary score (PCS) and the mental health summary score (MCS) can be derived from administering the tool. The scores on these two components are similar in magnitude and degree of change over time with values obtained using the longer version SF-36 questionnaire therefore making the SF-12 the instrument of choice where these 2 summary scores of health status are adequate.
Health related quality of life (HRQOL): Mood | 6 months
  HADS: The Hospital Anxiety and Depression Scale (HADS) is a popular and widely used well-validated measure of anxiety and depression in a general medical population of patients. A key advantage of the HADS is its simplicity, speed and ease of use. It assesses both anxiety and depression components which commonly co-exist using 7 domains on each component. Each domain has 4 descriptors with a score range 0-3 and a maximum total score of 21 possible for each component. Grade levels of mild, moderate and severe are defined by cut-off scores for each component.
Participant Satisfaction with telerehabilitation intervention | 6 months
  User satisfaction questionnaire will be administered following the intervention as a measure of acceptance and satisfaction with engaging in guided self-rehabilitation through the use of telerehabilitation technology. This will be administered in the post intervention assessment only.
  The user satisfaction questionnaire will be administered as part of the post intervention assessment to evaluate the views and opinions of the study participants with regards to using the Intendu Active Brain Trainer as part of their rehabilitation programme. This questionnaire has been developed for this study based on published evidence of the identified factors associated between telehealth and patient satisfaction.
Leisure Time Physical Activity | 6 months
  Leisure time physical activity behaviour will be evaluated by administering the Godin leisure time exercise questionnaire (Godin LTQ). This is a self-report paper based questionnaire that will be administered pre and post intervention.The Godin leisure time questionnaire is a simple 3 item tool that has well established validity and reliability for assessment of leisure time behaviour and offering a means of examining changes in behaviour following implementation of health intervention programmes.

CONTACTS AND LOCATIONS:
Locations (1):
- Castle Hill Hospital (Hull and east Yorkshire Hospitals NHS Trust), Cottingham, East Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No plans to share individual participant data